CLINICAL TRIAL: NCT05215327
Title: Comparison of High Dose vs. Standard Dose Influenza Vaccines in Lung Allograft Recipients
Brief Title: High vs. Standard Dose Influenza Vaccine in Lung Allograft Recipients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Northwestern University Feinberg School of Medicine (Other); University of Alabama at Birmingham (Other); Duke University (Other); University of Washington (Other); Emory University (Other); Baylor College of Medicine (Other); NYU Langone Health (Other)
Responsible Party: Principal Investigator, Natasha Halasa, Professor of Pediatric Infectious Diseases, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 212201
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Immunization; Infection; Transplantation Infection; Influenza
Keywords: Influenza; Vaccination; Immunization; Lung Transplantation; High Dose; Fluzone; Standard Dose; Influenza, Human; Communicable Diseases
MeSH Terms: conditions — Infections; Influenza, Human; Communicable Diseases | interventions — Influenza Vaccines; Fluzone High-Dose

STUDY DESIGN:
Intervention Model Description: The primary goal of this study is to compare influenza vaccine immunogenicity and safety between two doses of HD-QIV and two doses of SD-QIV in a population of lung transplant recipients. The study will be powered on a comparison of the primary immunogenicity outcome. A nominal level of α = 0.05 (two-sided) will be used to determine statistical significance
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study staff, and subjects will be blinded to which vaccine the subject will receive, except for an un-blinded vaccinator. This individual will not inform the study team or the subjects which vaccine they administered to the subject. The un-blinded vaccinator will not participate in any other study activities. If the study vaccine is provided in a blinded manner, then research staff will be able to administer the vaccine, and an un-blinded vaccinator will not be necessary. The pharmacy will be un-blinded and will have a record of which vaccine was given to each subject.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Two Doses High Dose Quadrivalent Inactivated Influenza Vaccine (Experimental): two doses of HD-QIV (0.7 mL; 60µg of each influenza antigen) 28-42 days apart
  Interventions: Biological: High Dose Quadrivalent Inactivated Influenza Vaccine
- Two Doses Standard Dose Quadrivalent Inactivated Influenza Vaccine (Experimental): receive two doses of SD-QIV (0.5 mL; 15µg of each influenza antigen) 28-42 days apart
  Interventions: Biological: Standard Dose Quadrivalent Inactivated Influenza Vaccine

INTERVENTIONS:
Biological: High Dose Quadrivalent Inactivated Influenza Vaccine — Fluzone High-Dose (Influenza Vaccine) for intramuscular injection is an inactivated influenza vaccine, prepared from influenza viruses propagated in embryonated chicken eggs. The virus-containing allantoic fluid is harvested and inactivated with formaldehyde. Influenza virus is concentrated and purified in a linear sucrose density gradient solution using a continuous flow centrifuge. The virus is then chemically disrupted using a non-ionic surfactant, octylphenol ethoxylate (Triton® X-100), producing a "split virus". The split virus is further purified and then suspended in sodium phosphatebuffered isotonic sodium chloride solution. The Fluzone High-Dose process uses an additional concentration factor after the ultrafiltration step in order to obtain a higher hemagglutinin (HA) antigen concentration.
  Other Names: Fluzone High Dose
  Arms: Two Doses High Dose Quadrivalent Inactivated Influenza Vaccine
Biological: Standard Dose Quadrivalent Inactivated Influenza Vaccine — Fluzone ® Quadrivalent is a vaccine indicated for active immunization for the prevention of influenza disease caused by two influenza A subtype viruses and two type B viruses contained in the vaccine.
  Other Names: Fluzone
  Arms: Two Doses Standard Dose Quadrivalent Inactivated Influenza Vaccine

SUMMARY:
Lung allograft recipients have a higher burden of influenza disease and greater associated morbidity and mortality compared with healthy controls. Induction and early maintenance immunosuppression is thought to impair immunogenicity to standard dose inactivated influenza vaccine. This early post-transplant period is when immunity is most desirable, since influenza disease during this time frame is associated with adverse consequences. Thus, strategies to reduce severe influenza disease in this highly susceptible population are critical. No trials in lung transplant recipients have evaluated two doses of HD-IIV within the same influenza season as a strategy to improve immunogenicity and durability of influenza prevention. Furthermore, no influenza vaccine trials have focused on enrollment of subjects at early post-transplant timepoints. Very few studies have been performed in solely lung allograft recipients. Immunosuppression intensity is highest in lung patients, thereby limiting comparisons to recipients of heart, liver, and kidney transplants. Therefore, studies to assess both HD-IIV and two-dose strategies in the same influenza season in post-lung transplant recipients are greatly needed.

The central hypothesis of our proposal is that lung allograft recipients who are 1-35 months post-transplant and receiving two doses of HD-quadrivalent inactivated influenza vaccine (QIV) will have higher HAI geometric mean titers (GMT) to influenza antigens compared to those receiving two doses of SD-QIV. To test this hypothesis and address the above critical knowledge gaps, we propose to conduct a phase II, multi-center, randomized, double-blind, controlled immunogenicity and safety trial comparing the administration of two doses of HD-QIV to two doses of SD-QIV in lung allograft recipients 1-35 months post-transplant. The results of this clinical trial will address significant knowledge gaps regarding influenza vaccine strategies (e.g., one vs. two doses and HD-QIV vs. SD-QIV) and immune responses in lung transplant recipients and will guide vaccine recommendations during the post-transplant period.

DETAILED DESCRIPTION:
Study Design: The proposed study is a phase II, multi-center, double-blind, randomized controlled immunogenicity and safety trial comparing two doses of HD-QIV to two doses of SD-QIV in lung allograft recipients.

1. Hypothesis 1: We hypothesize that lung allograft recipients 1-35 months post-transplant who receive two doses of HD-QIV will develop higher HAI GMTs to influenza antigens compared to lung allograft recipients receiving two doses of SD-QIV.

   Specific Aim 1: To compare the HAI GMTs to influenza antigens in lung allograft recipients after receiving either two doses of HD-QIV or two doses of SD-QIV.
2. Hypothesis 2: We hypothesize that administration of two doses of HD-QIV in lung transplant recipients will be well tolerated and the safety profile will be similar to two doses of SD-QIV with regard to solicited local and systemic side effects.

   Specific Aim 2: To compare the frequency and severity of solicited local and systemic adverse events in lung allograft recipients after receiving either two doses of HD-QIV or two doses of SD-QIV.
3. Hypothesis 3: We hypothesize that baseline immunophenotypic markers of exhaustion, immune senescence, and immune activation at the pre-vaccine timepoint will correlate with post-vaccine HAI titers.

Specific Aim 3: To define the relationship between baseline phenotypes of T- and B-cell subsets, T-cell activation and post-vaccination HAI titers among lung allograft recipients receiving either two doses of HD-QIV or two doses of SD-QIV.

Study Population: The study will enroll a total of approximately 270 subjects ≥16 years who have undergone lung transplantation within 1-35 months.

Study Enrollment: The enrollment period will be over a three-years. Subjects will be randomized into one of two groups. Group 1 will receive two doses of HD-QIV (0.7 mL; 60μg of each influenza antigen), whereas Group 2 will receive two doses of SD-QIV (0.5 mL; 15μg of each influenza antigen).

Influenza Surveillance: Active surveillance for influenza-like symptoms will begin when influenza season starts in each site's community, defined in previous trials as identification of at least two positive respiratory tests for influenza, with at least 10% of diagnostic tests positive during two consecutive weeks in the local clinical or research laboratory.41,42 Enrollment will continue during influenza season with nasal swabs obtained at all main visits to document the occurrence of influenza virus both prior to and after vaccination. During the influenza season, the study staff will attempt to do a weekly telephone and/or electronic communication with the participants to detect and document any influenza-like illness (ILI) and any specific COVID-19 like symptoms.

If subjects meet ILI criteria and/or any specific COVID-19 like symptoms (see below), an additional nasal swab will be collected*.

ILI criteria are met by occurrence of one of the conditions below:

* Fever: ≥38°C (100.4°F)
* Two or more of any of the following: respiratory symptoms (rhinorrhea, sinus congestion, post-nasal drip, shortness of breath, cough, wheezing, sputum production, sore throat, sneezing, watery eyes, ear pain, hoarseness); or systemic symptoms (myalgias, chills, chest pain, or headache); or new loss of taste or new loss of smell; or gastrointestinal symptoms (diarrhea or vomiting).

  * Per investigators' discretion at each individual site, a swab is not needed if there is a known non-respiratory cause of symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Lung allograft recipients
2. Age ≥16 years at time of enrollment
3. ≥1 month (30 days) and <36 months post-lung transplant
4. Anticipated to be available for duration of the study
5. Can be reached by telephone, email, or text message

Exclusion Criteria:

1. Recipient of multi-organ, extra-pulmonary, and/or hematopoietic stem cell transplant
2. Recipient of a re-do lung transplant
3. History of severe hypersensitivity to previous influenza vaccination or anaphylaxis to eggs/egg protein
4. History of Guillain-Barre syndrome
5. HIV positive patients, by history or documentation from previous test
6. History of known severe latex hypersensitivity
7. History of receiving the current season's influenza vaccine post-transplant prior to enrollment in the study
8. Pregnant female
9. Proven influenza disease after September 1st and before first study vaccine (patient can still receive the second influenza vaccination despite proven influenza disease once enrolled)
10. CMVIG/IVIG/SCIG receipt within 28 days of each vaccine
11. Receipt of rituximab or other B-cell depleting antibody (including proteasome inhibitors) therapy within 3-months of 1st study vaccine (Day 0).
12. Receipt of augmented T-cell depleting therapy within 3-months of 1st study vaccine (Day 0)
13. Investigator concern about study participation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Geometric Mean Titers of influenza vaccine antibodies. | Day 56 (post-vaccination)
  Antibody titers will be measured by hemagglutination inhibition assay.
The number of participants reporting solicited injection site reactions and systemic reactions. | Within 7 days post-vaccination
  Post-vaccination local adverse events (pain, tenderness, swelling/induration, erythema/redness, swelling/induration size, and erythema/redness size) and systemic adverse events (Fatigue/malaise, headache, nausea, body ache/myalgia (not at the injection site), general activity level, vomiting, and fever).

SECONDARY OUTCOMES:
Geometric Mean Titers Ratio of influenza vaccine antibodies (post-/pre-vaccination). | Day 56 (post-vaccination)
  Antibody titers will be measured by hemagglutination inhibition assay.
The number of participants achieving seroprotection and seroconversion for influenza virus. | Day 56 (post-vaccination)
  Antibody titers will be measured by hemagglutination inhibition assay. Seroconversion is defined as ≥ 4-fold rise in hemagglutination inhibition assay titers. Seroprotection is defined as ≥1:40 hemagglutination inhibition assay titer.

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Halasa, MD. MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No